CLINICAL TRIAL: NCT00744562
Title: A Phase 1 Dose Escalation Study of OMP-21M18 in Subjects With Solid Tumors
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: OncoMed Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Organization: Mereo BioPharma (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: M18-001
Record Dates: First submitted 2008-08-29; First posted 2008-09-01 (Estimated); Last update posted 2020-09-10 (Actual); Status verified 2020-09

CONDITIONS: Solid Tumors
Keywords: Phase 1,; dose escalation,; histologically; confirmed; malignancy; metastatic
MeSH Terms: conditions — Neoplasms; Neoplasm Metastasis | interventions — demcizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Open-label OMP-21M18 (Experimental)
  Interventions: Drug: OMP-21M18

INTERVENTIONS:
Drug: OMP-21M18 — 0.5, 1, 2.5, 5, and 10 mg/kg weekly until day 56. If patient has not progressed may continue with original dose administered every other week until progression

SUMMARY:
A phase 1 open-label dose escalation study of OMP-21M18 in subjects with previously treated solid tumour for which there is no remaining standard curative therapy and no therapy with a demonstrated survival benefit.

DETAILED DESCRIPTION:
This is an open-label Phase 1 dose escalation study of OMP-21M18 in subjects with previously treated solid tumors for which there is no remaining standard curative therapy and no therapy with a demonstrated survival benefit. Up to 30 subjects will be enrolled at up to 4 centers. Subjects will be assessed for safety, immunogenicity, pharmacokinetics, biomarkers, and efficacy. No formal interim analyses will be performed. Prior to enrollment, subjects will undergo screening to determine study eligibility. Upon enrollment, subjects will receive weekly intravenous (IV) infusions of OMP-21M18 for 9 weeks. After 9 weeks of treatment, subjects will be assessed for disease status. If there is no evidence of disease progression or if the tumor is smaller, then subjects may continue to receive IV infusions of OMP-21M18 every other week until disease progression.

Dose escalation will be conducted to determine the maximum tolerated dose (MTD). The dose levels of OMP 21M18 will be 0.5, 1.0, 2.5, 5, and 10 mg/kg administered IV weekly for 9 doses. No dose escalation or reduction will be allowed within a dose cohort. The dose may be administered at any time during the day. Three subjects will be treated at each dose level if no dose-limiting toxicities (DLTs) are observed. If 1 of 3 subjects experience a DLT, that dose level will be expanded to 6 subjects. If 2 or more subjects experience a DLT, no further subjects will be dosed at that level and 3 additional subjects will be added to the preceding dose cohort unless 6 subjects have already been treated at that dose level. Subjects will be assessed for DLTs from the time of the first dose through 7 days after administration of the 4th dose, but prior to administration of the 5th dose (i.e., Days 0-28). Dose escalation, if appropriate, will occur after all subjects in a cohort have completed their Day 28 DLT assessment.

ELIGIBILITY:
Inclusion Criteria:

1. Subjects must have a histologically confirmed malignancy that is metastatic or unresectable for which there is no remaining standard curative therapy and no therapy with a demonstrated survival benefit. In addition, subjects must have a tumor that is at least 2 x 2 cm and is radiographically apparent on CT or MRI.
2. Subjects must have received their last chemotherapy, biologic, or investigational therapy at least 4 weeks prior to enrollment, 6 weeks if the last regimen included BCNU or mitomycin C.
3. Age >21 years
4. ECOG performance status <2
5. Life expectancy of more than 3 months
6. Subjects must have normal organ and marrow function as defined below:

   * Leukocytes >3000/mL
   * Absolute neutrophil count >1000/mL
   * Hemoglobin >9.0 g/dL
   * Platelets >100,000/mL
   * Total bilirubin <1.5 X institutional upper limit of normal (ULN)
   * AST (SGOT) and ALT (SGPT) <2.5 X institutional ULN
   * PT and PTT within institutional ULN
   * Creatinine <1.5 X institutional ULN OR
   * Creatinine clearance >60 mL/min/1.73 m2 for subjects with creatinine levels above institutional normal
7. Women of childbearing potential must have had a prior hysterectomy or have a negative serum pregnancy test and be using adequate contraception prior to study entry and must agree to use adequate contraception from study entry through at least 6 months after discontinuation of study drug. Men must also agree to use adequate contraception (hormonal or barrier method of birth control; abstinence) prior to study entry and from study entry through at least 6 months after discontinuation of study drug.

Exclusion Criteria:

1. Subjects receiving any other investigational agents
2. Subjects with known brain metastases, uncontrolled seizure disorder, or active neurologic disease
3. History of a significant allergic reaction attributed to humanized or human monoclonal antibody therapy
4. Significant intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements
5. Pregnant women or nursing women
6. Subjects with known HIV infection
7. Known bleeding disorder or coagulopathy
8. Subjects receiving heparin, warfarin, or other similar anticoagulants. Note: Subjects may be receiving low-dose aspirin and/or non-steroidal anti-inflammatory agents.
9. Subjects with known clinically significant gastrointestinal disease including, but not limited to, inflammatory bowel disease

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 42 (Actual)
Dates: Start 2008-08; Primary Completion 2011-11 (Actual); Study Completion 2012-01 (Actual)

PRIMARY OUTCOMES:
To determine the safety of OMP-21M18 in subjects with previously treated solid tumors | continuous

SECONDARY OUTCOMES:
To determine the pharmacokinetics of OMP-21M18 in subjects with previously treated solid tumors | First 8 doses and following treatment termination

CONTACTS AND LOCATIONS:
Locations (3):
- United States (3):
  - California Cancer Care, Greenbrae, California
  - Stanford University, Stanford, California
  - University of Michigan Comprehensive Cancer Center, Ann Arbor, Michigan